CLINICAL TRIAL: NCT05512481
Title: A Phase 2 Clinical Trial of Neoadjuvant Camrelizumab Plus Apatinib and Temozolomide in High Risk Clinical Stage Ⅱ-Ⅲ Acral Melanoma
Brief Title: Camrelizumab Plus Apatinib and Temozolomide as Neoadjuvant in High Risk Acral Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Jun Guo, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-MM-Ⅱ-003
Record Dates: First submitted 2022-08-21; First posted 2022-08-23 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Melanoma; Acral Melanoma; Temozolomide; Apatinib; Camrelizumab; Neoadjuvant; Pathological Response
Keywords: Acral Melanoma; Immune Checkpoint Inhibitors; Protein Kinase Inhibitors; Antineoplastic Agents, Alkylating
MeSH Terms: conditions — Melanoma | interventions — camrelizumab; apatinib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant/adjuvant therapy (Experimental): Drug: Camrelizumab
  Drug: Apatinib mesylate
  Drug: Temozolomide Injection
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — NEOADJUVANT:
  All participants will receive neoadjuvant therapy with combination of Camrelizumab、Apatinib and Temozolomide for 2 cycle；
  SURGERY: All participants will have melanoma surgery after 2 cycles of treatment
  ADJUVANT: Participants will receive Camrelizumab every 3 weeks for 1 year
  Other Names: Apatinib; Temozolomide

SUMMARY:
Neoadjuvant therapy is feasible in stage Ⅱ-Ⅲ melanoma, Carrelizumab combined with apatinib and temozolomide has synergistic antitumor effects and may improve pathological response.

DETAILED DESCRIPTION:
Patients with resectable melanoma can benefit from neoadjuvant therapy, including improved surgical outcomes, precise management of patients based on neoadjuvant response, and analysis of resistance mechanisms through histological sections for subsequent treatment. At present, there have been a number of clinical trials exploring the effect of neoadjuvant regimens for melanoma, and some published results have shown that neoadjuvant therapy can lead to a higher pathological response rate, thereby improving the RFS of patients.

In the past, this site has carried out a clinical study of Camrelizumab combined with Apatinib and Temozolomide for first-line treatment of unresectable acral melanoma, with a high preliminary clinical response rate and safety. Based on this, this study intends to evaluate the neoadjuvant treatment of completely resectable melanoma with Camrelizumab combined with Apatinib and Temozolomide in patients with stage III and IIB, IIC high-risk melanoma. To comprehensively evaluate the short-term and long-term benefits of neoadjuvant therapy and provide an important reference for neoadjuvant treatment strategies in the acral melanoma population.

ELIGIBILITY:
Inclusion Criteria:

1. age:18-75 years, male or female.
2. Histopathologically confirmed acral melanoma (stage Ⅱ/Ⅲ).
3. Has not received any systematic anti-tumor drug treatment.
4. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.
5. ECOG 0-1.
6. Adequate organ function.
7. Life expectancy of greater than 12 weeks.
8. Patient has given written informed consent.

Exclusion Criteria:

1. Patients who have or are currently undergoing additional chemotherapy, radiation therapy, targeted therapy or immunotherapy.
2. Known history of hypersensitivity to any component of apatinib, temozolomide, Camrelizumab.
3. Subjects before or at the same time with other malignant tumors (except which has cured skin basal cell carcinoma and cervical carcinoma in situ);
4. Subjects with any active autoimmune disease or history of autoimmune disease
5. Patients with any unstable systemic disease, including but not limited to: serious infection, uncontrolled diabetes, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, myocardial infarction, congestive heart failure, serious cardiac arrhythmia requiring medication, hepatic, renal or metabolic disease;
6. Received a live vaccine within 4 weeks of the first dose of study medication.
7. Pregnancy or breast feeding.
8. Decision of unsuitableness by principal investigator or physician-in charge.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | Week 8-12
  The primary endpoint is the pathological response rate at surgery after neoadjuvant study treatment.
  The pathological response is categorised thus:
  Complete pathological response (pCR) - 0% viable tumour cells in the surgical specimen Near complete pathological response - (near pCR) - <10% viable tumour Partial pathological response (pPR) - 10%-50% viable tumour No pathological response (pNR) - >50% viable tumour

SECONDARY OUTCOMES:
Objective Response Rate | Months 0-6
  Disease Response as assessed by RECIST 1.1 and mRECIST
Recurrence-free survival | 1year,2year
  The proportion of patients with an histologically confirmed diagnosis of disease recurrence (local, regional, and distant), as detected by the patient, on physical examination or during imaging surveillance, or death from any cause.
Overall survival | 10 years
  The proportion of participants deceased from any cause.
Safety and tolerability of neoadjuvant and adjuvant treatment and surgical procedures. | 90 days from last dose of study treatment
  The proportion of patients with adverse events as described in CTCAE version 5.0
Patient reported quality of life | 90 days from last dose of study treatment
  The individual, summary and composite scores obtained from the validated EUROQOL QLQ-C30 questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Guo, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No